CLINICAL TRIAL: NCT01513629
Title: Structural Connectivity as Imaging Endophenotypes of Autism Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Statistical Center, NTUHCTC, Wen-Yih Isaac Tseng, MD, PhD, National Taiwan University Hospital
Other Study IDs: 201006032R
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism spectrum disorders; structural connectivity; diffusion spectrum imaging; sibling; endophenotype
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Autism spectrum disorders (ASD) is a highly hereditary neuropsychiatric disorder. In children and adolescents worldwide, the prevalence of ASD is estimated at 0.6%. Understanding the biological mechanism of this disorder could potentially facilitate prompt, accurate and personalized therapy. The dysfunction of fronto-temporal circuitry may explain language impairment in ASD. In addition, pieces of evidence suggest that the abnormality of the cortico-striato-thalamic circuitry might be related to social deficits. However, very little is known how changes in these two circuitries are related to variation in genotypes. Previous reports on ASD using magnetic resonance imaging (MRI) have demonstrated alteration of brain structure. Recent advance in neuroimaging has shown that structural connectivity of a specific circuitry is superior to regional analysis in terms of higher penetrance of genetic effects and better account for behavioral variance. Therefore, it is plausible that connectivity imaging may serve as effective endophenotypes that link clinical manifestation (phenotypes) and the biological variables (genotypes). In the past five years, our lab has established world leading diffusion spectrum imaging techniques, and applied the techniques to clinical studies on ASD, schizophrenia, stroke and epilepsy. The clinical experience and technical strengths provide a strong basis for us to extend to imaging genetics, aiming to determine effective endophenotypes of ASD. Therefore, the goal of this project is to validate structural connectivity of fronto-temporal and cortico-striato-thalamic circuitries as effective imaging endophenotypes of ASD. Specifically, the investigators will achieve the goal through a series of validation. First, the investigators will demonstrate that structural connectivities in the two targeted circuitries are indeed different among groups of patients with ASD, unaffected siblings, and neurotypicals. Second, the investigators will demonstrate in neurotypicals and unaffected siblings that the altered structural connectivities related to social and language impairments are indeed different in carriers of risk genes, i.e. CNTNAP2 and SLC25A12, respectively. Last, the investigators will demonstrate in all participants that the altered structural connectivities are associated with the corresponding behavioral variances in social and language function. This two-year project is a cohort study consisting of three groups, namely patient, unaffected siblings, and control groups matched in age, gender and handedness. The patient and sibling groups consist of 20 boys each, age 10-15 years old, and the control group consists of 40 boys. The examination includes behavior assessment (IQ test, neuropsychological and clinical assessment), MRI study (structure MRI and diffusion spectrum imaging for structural connectivity) and genome scan(specifically candidate genes related to language function, i.e. SLC25A12, and to social function, i.e. CNTNAP2). In conclusion, this is the first cohort project on imaging genetics in Taiwan. The success of this project will facilitate the progress of translational neuroscience in Taiwan. The methodology of validating endophenotype will be readily extended to other psychiatric diseases.

ELIGIBILITY:
Inclusion Criteria:

* 20 males, right handed, age 10-15 years old. Diagnosis of high-functioning autism is made according to the DSM-IV and ICD-10 criteria by senior child psychiatrists experienced in autism assessments and treatments. The patients should have full-scale IQ ≧ 80 and no comorbid diseases.
* 20 unaffected (discordant) male siblings of patients with high-functioning autism
* 40 healthy school boys without any psychiatric disorders in the 1st and 2nd degree relatives. The patient group (N=20) and a neurotypical group (N=20) are matched in age,gender and handedness. The family group (N=20) and another neurotypical group (N=20) are matched in age, gender and handedness.

Exclusion Criteria:

* full-scale IQ < 80 and with comorbid diseases
* large imaging motion artifact

Ages: 10 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: High-functioning autism group,family group, and neurotypical group
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2012-09-30 (Actual); Study Completion 2012-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Yih I Tseng, MD, PhD, Principal Investigator — Center for Optoelectronic Biomedicine, National Taiwan University College of Medicine
Locations (1):
- Center for Optoelectronic Biomedicine, National Taiwan University College of Medicine, Taipei, Taiwan